CLINICAL TRIAL: NCT04379596
Title: A Phase 1b/2 Multicenter, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of Trastuzumab Deruxtecan (T-DXd) Monotherapy and Combinations in Adult Participants With HER2-expressing Gastric Cancer (DESTINY-Gastric-03)
Brief Title: Ph1b/2 Study of the Safety and Efficacy of T-DXd Combinations in Advanced HER2-expressing Gastric Cancer (DESTINY-Gastric03)
Acronym: DG-03
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D967LC00001; 2019-004483-22 (EudraCT Number)
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Esophageal Cancer; Carcinoma; HER2; Trastuzumab; Deruxtecan; T-DXd; DS-8201a; Gastroesophageal Cancer; Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Carcinoma; Adenocarcinoma | interventions — Fluorouracil; Capecitabine; durvalumab; Oxaliplatin; Trastuzumab; trastuzumab deruxtecan; Cisplatin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: The study will consist of 2 phases: a dose escalation phase (Part 1) and dose expansion phases (Part 2, Part 3, Part 4 and Part 5). Part 1 will enroll HER2-overexpressing (IHC 3+ or IHC 2+/ISH+), previously treated gastric, gastro-esophageal junction (GEJ) or esophageal cancer patients, and Part 2 will enroll HER2-overexpressing patients who have not received prior treatment for metastatic or unresectable disease. Part 3, Part 4 and Part 5 will enroll HER2-expressing patients who have not received prior treatment for metastatic or unresectable disease.
  In addition to safety and tolerability, this study will also assess ORR, DoR, DCR, OS, PFS and other measures of antitumor activity among treatment groups. Tumor evaluation using RECIST v1.1 will be conducted at screening and every 6 weeks until RECIST 1.1 objective disease progression or withdrawal of consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Arm 1A (Experimental): T-DXd and 5-fluorouracil (5-FU)
  Interventions: Drug: Fluorouracil (5-FU); Drug: Trastuzumab deruxtecan
- Arm 1B (Experimental): T-DXd and capecitabine
  Interventions: Drug: Capecitabine; Drug: Trastuzumab deruxtecan
- Arm 1C (Experimental): T-DXd and durvalumab
  Interventions: Biological: Durvalumab; Drug: Trastuzumab deruxtecan
- Arm 1D(b) (Experimental): T-DXd, capecitabine, and oxaliplatin
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Trastuzumab deruxtecan
- Arm 1E(a) (Experimental): T-DXd, 5-FU, and durvalumab
  Interventions: Drug: Fluorouracil (5-FU); Biological: Durvalumab; Drug: Trastuzumab deruxtecan
- Arm 1E(b) (Experimental): T-DXd, capecitabine, and durvalumab
  Interventions: Drug: Capecitabine; Biological: Durvalumab; Drug: Trastuzumab deruxtecan
- Arm 2A (Active Comparator): Trastuzumab, 5-FU or capecitabine, and cisplatin or oxaliplatin
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Oxaliplatin; Biological: Trastuzumab; Drug: Cisplatin
- Arm 2B (Experimental): T-DXd monotherapy
  Interventions: Drug: Trastuzumab deruxtecan
- Arm 2C (Experimental): T-DXd, 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan
- Arm 2D (Experimental): T-DXd, pembrolizumab and 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan; Biological: Pembrolizumab
- Arm 2E (Experimental): T-DXd and pembrolizumab
  Interventions: Drug: Trastuzumab deruxtecan; Biological: Pembrolizumab
- Arm 2F (Experimental): T-DXd, pembrolizumab and 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan; Biological: Pembrolizumab
- Arm 3A (Experimental): T-DXd, Volrustomig and 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan; Biological: Volrustomig
- Arm 3B (Experimental): T-DXd, Volrustomig and 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan; Biological: Volrustomig
- Arm 4A (Experimental): T-DXd, Rilvegostomig and 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan; Biological: Rilvegostomig
- Arm 4B (Experimental): T-DXd, Rilvegostomig and 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan; Biological: Rilvegostomig
- Part 5 Main Cohort (Experimental): T-DXd, Volrustomig and 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan; Biological: Volrustomig
- Part 5 Cohort 2 (Experimental): T-DXd, Volrustomig and 5-FU or capecitabine
  Interventions: Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Trastuzumab deruxtecan; Biological: Volrustomig

INTERVENTIONS:
Drug: Fluorouracil (5-FU) — 5-FU: administered as an IV infusion
  Arms: Arm 1A; Arm 1E(a); Arm 2A; Arm 2C; Arm 2D; Arm 2F; Arm 3A; Arm 3B; Arm 4A; Arm 4B; Part 5 Cohort 2; Part 5 Main Cohort
Drug: Capecitabine — Capecitabine: administered orally
  Arms: Arm 1B; Arm 1D(b); Arm 1E(b); Arm 2A; Arm 2C; Arm 2D; Arm 2F; Arm 3A; Arm 3B; Arm 4A; Arm 4B; Part 5 Cohort 2; Part 5 Main Cohort
Biological: Durvalumab — Durvalumab: administered as an IV infusion
  Other Names: MEDI4736
  Arms: Arm 1C; Arm 1E(a); Arm 1E(b)
Drug: Oxaliplatin — Oxaliplatin: administered as an IV infusion
  Arms: Arm 1D(b); Arm 2A
Biological: Trastuzumab — Trastuzumab: administered as an IV infusion
  Arms: Arm 2A
Drug: Trastuzumab deruxtecan — T-DXd: administered as an IV infusion
  Other Names: DS-8201a, Enhertu
  Arms: Arm 1A; Arm 1B; Arm 1C; Arm 1D(b); Arm 1E(a); Arm 1E(b); Arm 2B; Arm 2C; Arm 2D; Arm 2E; Arm 2F; Arm 3A; Arm 3B; Arm 4A; Arm 4B; Part 5 Cohort 2; Part 5 Main Cohort
Drug: Cisplatin — Cisplatin: administered as an IV infusion
  Arms: Arm 2A
Biological: Pembrolizumab — Pembrolizumab: administered as an IV infusion
  Arms: Arm 2D; Arm 2E; Arm 2F
Biological: Volrustomig — Volrustomig: administered as an IV infusion
  Other Names: MEDI5752
  Arms: Arm 3A; Arm 3B; Part 5 Cohort 2; Part 5 Main Cohort
Biological: Rilvegostomig — Rilvegostomig: administered as an IV infusion
  Other Names: AZD2936
  Arms: Arm 4A; Arm 4B

SUMMARY:
DESTINY-Gastric03 will investigate the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary antitumor activity of trastuzumab deruxtecan (T-DXd) alone or in combination with chemotherapy and/or immunotherapy in HER2-expressing advanced/metastatic gastric/gastroesophageal junction (GEJ) and esophageal adenocarcinoma patients.

Study hypotheses: Combination of T-DXd with cytotoxic chemotherapy and/or immunotherapy administered to subjects at the recommended phase 2 dose will show manageable safety and tolerability and preliminary anti-tumor efficacy so as to permit further clinical testing. T-DXd in combination with cytotoxic chemotherapy or immune checkpoint inhibitor administered to HER2-expressing gastric, GEJ and esophageal cancer patients who have not received prior treatment for advanced/metastatic disease will show preliminary evidence of anti-tumour activity and the potential to become a therapeutic option for this patient population.

ELIGIBILITY:
Inclusion criteria:

1. Male and female participants must be at least 18 years of age. Other age restrictions may apply as per local regulations
2. Disease Characteristics:

   1. Locally advanced, unresectable, or metastatic disease based on most recent imaging
   2. For Part 1, 2, 3a, 4a pathologically documented adenocarcinoma of the stomach/GEJ/esophagus, HER2-positive (IHC 3+ or IHC 2+/ISH+) based on local tissue testing results
   3. For Part 3b,4b and Part 5, pathologically documented adenocarcinoma of the stomach/GEJ/esophagus, HER2-low (IHC 2+/ISH-negative or IHC 1+) based on local tissue testing results
3. For Part 1, progression on or after at least one prior trastuzumabcontaining regimen For Part 2, Part 3, Part 4 and Part 5, previously untreated for unresectable or metastatic adenocarcinoma of the stomach/GEJ/ esophagus with with HER2-positive (Part 2 and Part 3 [Arm 3A] and Part 4 [Arm 4A]) or HER2-low (Part 3 [Arm 3B], Part 4 [Arm 4B] and Part 5)) status
4. Has measurable target disease assessed by the Investigator based on RECIST version 1.1
5. Has protocol defined adequate bone marrow and organ function including cardiac, renal and hepatic function
6. If of reproductive potential, agrees to use a highly effective form of contraception or avoid intercourse during and upon completion of the study.

Exclusion criteria:

1. Part 1 to 4: History of active primary immunodeficiency, known HIV, active chronic, or past hepatitis B infection, or hepatitis C infection. Part 5: evidence of active, uncontroled HIV, HBV or HCV infection.
2. Uncontrolled intercurrent illness.
3. History of non-infectious pneumonitis/ILD, current ILD, or where suspected ILD that cannot be ruled out by imaging at screening.
4. Lung-specific intercurrent clinically significant severe illnesses.
5. Uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals.
6. Pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART).
7. Has spinal cord compression or clinically active central nervous system metastases.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Occurrence of adverse events (AEs) and serious adverse events (SAEs), graded according to NCI CTCAE v5.0 | Safety will be assessed up to the follow-up period, approximately 24 months.
  Occurrence of AEs and SAEs graded according to NCI CTCAE v5.0
Part 1: Ocurrence of dose-limiting toxicities (DLTs) | Safety will be assessed up to the follow-up period, approximately 24 months.
  Occurrence of dose limiting toxicities
Part 1: Changes from baseline in laboratory parameters | Safety will be assessed up to the follow-up period, approximately 24 months.
  Changes in laboratory parameters (every in appropriate units) compared to baseline results.
Part 1: Changes from baseline in vital signs | Safety will be assessed up to the follow-up period, approximately 24 months.
  Changes in vital signs results compared to baseline results.
Part 1: Changes from baseline in electrocardiogram (ECG) results | Safety will be assessed up to the follow-up period, approximately 24 months.
  Changes in ECG results compared to baseline results.
Part 2, Part 3, Part 4 and Part 5: Endpoint assessed by Investigator per RECIST v1.1: Confirmed Objective Response Rate (ORR) | (Endpoint: ORR) Efficacy will be assessed at an average of approximately 12 months
  Confirmed ORR per RECIST 1.1 is the percentage of patients with Complete Response or Partial Response that is subsequently confirmed.

SECONDARY OUTCOMES:
Part 1: Objective Response Rate (ORR) | Efficacy will be assessed at an average of approximately 12 months
  Confirmed ORR per RECIST 1.1 is the percentage of patients with Complete Response or Partial Response that is subsequently confirmed.
Part 2, Part 3, Part 4 and Part 5: Occurrence of adverse events (AEs) and serious adverse events (SAEs) | Safety will be assessed up to follow-up period, approximately 24 months
  Occurrence of AEs and SAEs graded according to NCI CTCAE v5.0
Part 2, Part 3, Part 4 and Part 5: Changes from baseline in laboratory parameters | Safety will be assessed up to follow-up period, approximately 24 months
  Changes in laboratory parameters (every in appropriate units) compared to baseline results.
Part 2, Part 3, Part 4 and Part 5: Changes from baseline in vital signs | Safety will be assessed up to follow-up period, approximately 24 months
  Changes in vital signs results compared to baseline results.
Part 2, Part 3 , Part 4 and Part 5: Changes from baseline in body weight | Safety will be assessed up to follow-up period, approximately 24 months
  Changes in body weight in kilograms compared to baseline results.
Part 2, Part 3, Part 4 and Part 5: Changes from baseline in electrocardiogram (ECG) results | Safety will be assessed up to follow-up period, approximately 24 months
  Changes in ECG results compared to baseline results.
Duration of Response (DoR) | Until progression or death, efficacy (DoR) will be assessed up to approximately 24 months
  DOR is defined as the time from the date of first documented response until the date of documented progression or death
Disease Control Rate (DCR) | Efficacy will be assessed at an average of approximately 12 months
  DCR is the percentage of subjects who have a best overall response of complete response (CR) or partial response (PR) or stable disease (SD)
Progression Free Survival (PFS) | Until progression or death, efficacy (PFS) will be assessed up to approximately 24 months
  PFS is the time from date of first dose until the date of objective disease progression or death
Overall survival (OS) | Until death, efficacy (OS) will be assessed up to approximately 24 months
  OS is the time from date of first dose until death due to any cause
Serum concentration of T-DXd, total anti-HER2 antibody, and MAAA-1181a in all arms | While on study drug up to study completion, approximately 24 months
  Individual participant data and descriptive statistics will be provided for serum concentration data at each time point for each dose level for T-DXd, total anti-HER2 antibody, MAAA-1181a
Serum concentration of durvalumab in study arms including T-DXd in combination with durvalumab | While on study drug up to study completion, approximately 24 months
  Individual participant data and descriptive statistics will be provided for serum concentration data at each time point for durvalumab.
Presence of ADAs for T-DXD, durvalumab, volrustomig and rilvegostomig (in study arms including T-DXd and durvalumab, and T-DXd and volrustomig, and T-DXd and rilvegostomig respectively) | While on study drug up to study completion, approximately 24 months
  Individual participant data and descriptive statistics will be provided for data at each time point for each dose level for T-DXd and durvalumab.
Serum concentrations of volrustomig and rilvegostomig in study arms including T-DXd in combination with volrustomig and T-DXd in combination with rilvegostomig | While on study drug up to study completion, approximately 24 months
  Individual participant data and descriptive statistics will be provided for data at each time point for rilvegostomig and volrustomig
Comparison of ORR | While on study drug up to study completion, approximately 24 months
  Comparison of objective response rate between participants using local HER2 test results and central HER2 test results from tumor samples with evaluable results
Comparison of DCR | While on study drug up to study completion, approximately 24 months
  Comparison of disease control rate between participants using local HER2 test results and central HER2 test results from tumor samples with evaluable results
Comparison of DoR | While on study drug up to study completion, approximately 24 months
  Comparison of duration of response between participants using local HER2 test results and central HER2 test results from tumor samples with evaluable results
Comparison of PFS | While on study drug up to study completion, approximately 24 months
  Comparison of progression-free survival between participants using local HER2 test results and central HER2 test results from tumor samples with evaluable results
Comparison of OS | While on study drug up to study completion, approximately 24 months
  Comparison of overall survival between participants using local HER2 test results and central HER2 test results from tumor samples with evaluable results

CONTACTS AND LOCATIONS:
Locations (77):
- United States (9):
  - Research Site, Santa Monica, California
  - Research Site, Westwood, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Brazil (9):
  - Research Site, Florianópolis
  - Research Site, Londrina
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, São Jose Do Rio Preto
  - Research Site, São Paulo
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (11):
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xiamen
  - Research Site, Zhengzhou
- Germany (5):
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Mannheim
  - Research Site, München
- Italy (5):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Verona
- Japan (4):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kita-gun
  - Research Site, Ota-shi
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Utrecht
- Poland (8):
  - Research Site, Gdansk
  - Research Site, Konin
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- Russia (4):
  - Research Site, Kostroma
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Santander
  - Research Site, Seville
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Dundee
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: ICF
Time Frame: Study start to completion date
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool .
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
  For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home